CLINICAL TRIAL: NCT05879939
Title: Transcutaneous Repetitive Phrenic Nerve Stimulation in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Sung Eun Hyun, Assistant professor (MD, PhD), Seoul National University Hospital
Other Study IDs: 2022R1F1A1071488
Record Dates: First submitted 2023-03-23; First posted 2023-05-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Electrical Stimulation; Phrenic Nerve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transcutaneous, repetitive phrenic nerve electrical stimulation — Phrenic nerve electrical stimulation with different stimulation intensity and frequency

SUMMARY:
The goal of this observational study is to characterize the standardized stimulation parameter for noninvasive, transcutaneous, repetitive phrenic nerve electrical stimulation.

The main questions it aims to answer are:

* Is the phrenic nerve repetitive electrical stimulation test feasible for use as non-invasive transcutaneous electrical stimulation?
* What is the most optimal stimulation parameters for repetitive phrenic nerve electrical stimulation in healthy adult populations in terms of effective and safe activation of diaphragm?

ELIGIBILITY:
Inclusion Criteria:

* Koreans who speak Korean as their mother tongue, aged 19 or older and younger than 40.
* Those who understood the purpose and procedure of this study and voluntarily participated with consent.

Exclusion Criteria:

1. - Those who have any neuromuscular disease.

   - Those whom abnormal findings are observed on a neurological examination. e.g.) Cases with abnormal findings in peripheral motor nerve (median nerve) and sensory nerve (sural nerve) conduction studies performed in screening.

   e.g.) People who have been diagnosed with a neuromuscular junctional diseases such as myasthenia gravis or receiving related treatment.
2. In the case of implantable electronic medical devices such as pacemakers, implantable cardioverter defibrillators (ICDs), and spinal cord stimulation devices.
3. Those who have any history of radiation therapy or chemotherapy for cancer within a year.
4. People who have a history of cardiovascular or cerebrovascular disease or lung disease within 6 months.
5. Those who have been diagnosed with a psychiatric/neurological problem or taking related medications that may affect electrophysiological study.
6. Those who are pregnant or may be pregnant.
7. Those who are judged to lack the cognitive ability to understand the explanation of the purpose and procedure of this study.
8. Those whom the researchers judge for other reasons to be inappropriate to participate in this study.

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult population who have read the recruitment announcement, voluntarily expressed their intention to participate, and have met the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Phrenic nerve compound muscle action potential (CMAP) amplitude (mV) | Baseline
  ∙ CMAP Amplitude (mV)
∙ Phrenic nerve compound muscle action potential (CMAP) duration (ms) | Baseline
  ∙ CMAP duration (ms)
∙ Phrenic nerve compound muscle action potential (CMAP) area (mV∙ms) | Baseline
  ∙ CMAP area (mV∙ms)

SECONDARY OUTCOMES:
Respiratory function | Baseline
  ∙ Maximum inspiratory pressure (MIP)
Diaphragmatic function | Baseline
  ∙ Baseline diaphragm thickness
Diaphragmatic function | Baseline
  ∙ Diaphragm thickening fraction percent: the difference between diaphragm thickness at the end of inspiration (DTi) and at the end of expiration (DTe) divided by DTe × 100
Pain during phrenic stimulation | Baseline
  ∙ Numeric rating scale (range: 0~10): This scale ranges from 0 to 10 points, with higher scores indicating more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Eun Hyun, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided